CLINICAL TRIAL: NCT05547412
Title: Validation of Velocity Curvature Index as a Diagnostic Biomarker Tool for Assessment of Large Vessel Stroke
Acronym: VOICE
Status: Terminated | Type: Observational
Why Stopped: enrollment, administrative/finance
Sponsor: NovaSignal Corp. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: NA-01STR-03; U44NS109952 (NIH)
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Results first posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-03

CONDITIONS: Stroke; Acute Ischemic Stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (6):
- Cohort X: Phase 0 will include up to 20 subjects in Cohort X (TCD). This phase is for training and feasibility purposes only and data collected will not be used in the final analysis.
  Interventions: Device: NovaGuide 2 Intelligent Ultrasound System
- Cohort Y: Phase 0 will include up to 20 subjects in Cohort Y (No TCD). This phase is for training and feasibility purposes only and data collected will not be used in the final analysis.
- Cohort A: Both Phase 1 and Phase 2 of the study will enroll Cohort A (LVO TCD). Cohort A will enroll 54 subjects in Phase 1 and 156 subjects in Phase 2
  Interventions: Device: NovaGuide 2 Intelligent Ultrasound System
- Cohort B: Both Phase 1 and Phase 2 of the study will enroll Cohort B (Non-LVO TCD). Cohort B will enroll 54 subjects in Phase 1 and 156 subjects in Phase 2
  Interventions: Device: NovaGuide 2 Intelligent Ultrasound System
- Cohort C: Both Phase 1 and Phase 2 of the study will enroll Cohort C (LVO No-TCD). Cohort C will enroll 54 subjects in Phase 1 and 156 subjects in Phase 2
- Cohort D: Both Phase 1 and Phase 2 of the study will enroll Cohort D (Non-LVO No-TCD). Cohort D will enroll 54 subjects in Phase 1 and 156 subjects in Phase 2

INTERVENTIONS:
Device: NovaGuide 2 Intelligent Ultrasound System — The NovaGuide 2 Intelligent Ultrasound system is an adjunctive mobile, non-invasive, non-ionizing radiation transcranial Doppler (TCD) diagnostic ultrasound system. The system contains a transcranial doppler ultrasound equipment combined with robotic mechanisms used to position ultrasound probes, which assist the user in the acquisition of cerebral blood flow velocity (CBFV) data via a patient's temporal acoustic windows.
  Groups: Cohort A; Cohort B; Cohort X

SUMMARY:
This study is a multi-center, multi-phase, multi-cohort, prospective, randomized, open, blinded endpoint (PROBE), non-significant risk (NSR) device study including up to 420 evaluable subjects measured with the study device(s) and up to 40 non-evaluable subjects for the training phase.

DETAILED DESCRIPTION:
The purpose of this study is to collect robust data from NovaGuide 2 Intelligent Ultrasound System to validate the Velocity Curvature Index (VCI) as a diagnostic biomarker tool to drive clinical decision making for assessing cerebral vascular occlusions confirmed by standard of care Computed Tomography Angiography (CTA) imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Subject aged 18 years and older referred for evaluation of possible stroke.
2. Subject receives Computed Tomography Angiography (CTA) imaging for the assessment of stroke.
3. Subject or Legally Authorized Representative has the ability to provide informed consent and comply with the protocol.

Exclusion Criteria:

1. Head CT findings consistent with acute primary intracranial hemorrhage (ICH), etc.
2. Subjects with occlusions in the distal or posterior circulation arteries.
3. Subjects who underwent partial or full craniotomy
4. Additional intracranial pathologies present (tumor, hydrocephalus, etc.)
5. Anticipated insufficient time to acquire a complete TCD scan as described by the protocol
6. Subjects who have a physical limitation preventing placement of the system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be enrolled from Stroke centers in the U.S.
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hamilton, Ph.D., Principal Investigator — NovaSignal Corp.
Locations (1):
- CHI Memorial Hospital, Chattanooga, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hastrup S, Damgaard D, Johnsen SP, Andersen G. Prehospital Acute Stroke Severity Scale to Predict Large Artery Occlusion: Design and Comparison With Other Scales. Stroke. 2016 Jul;47(7):1772-6. doi: 10.1161/STROKEAHA.115.012482. Epub 2016 Jun 7. PMID 27272487
- [Background] Smith EE, Kent DM, Bulsara KR, Leung LY, Lichtman JH, Reeves MJ, Towfighi A, Whiteley WN, Zahuranec DB; American Heart Association Stroke Council. Accuracy of Prediction Instruments for Diagnosing Large Vessel Occlusion in Individuals With Suspected Stroke: A Systematic Review for the 2018 Guidelines for the Early Management of Patients With Acute Ischemic Stroke. Stroke. 2018 Mar;49(3):e111-e122. doi: 10.1161/STR.0000000000000160. Epub 2018 Jan 24. PMID 29367333
- [Background] Thorpe SG, Thibeault CM, Wilk SJ, O'Brien M, Canac N, Ranjbaran M, Devlin C, Devlin T, Hamilton RB. Velocity Curvature Index: a Novel Diagnostic Biomarker for Large Vessel Occlusion. Transl Stroke Res. 2019 Oct;10(5):475-484. doi: 10.1007/s12975-018-0667-2. Epub 2018 Oct 6. PMID 30293170
- [Background] Thorpe SG, Thibeault CM, Canac N, Wilk SJ, Devlin T, Hamilton RB. Decision Criteria for Large Vessel Occlusion Using Transcranial Doppler Waveform Morphology. Front Neurol. 2018 Oct 17;9:847. doi: 10.3389/fneur.2018.00847. eCollection 2018. PMID 30386287
- [Background] Jalaleddini K, Canac N, Thorpe SG, O'Brien MJ, Ranjbaran M, Delay B, Dorn AY, Scalzo F, Thibeault CM, Wilk SJ, Hamilton RB. Objective Assessment of Beat Quality in Transcranial Doppler Measurement of Blood Flow Velocity in Cerebral Arteries. IEEE Trans Biomed Eng. 2020 Mar;67(3):883-892. doi: 10.1109/TBME.2019.2923146. Epub 2019 Jun 17. PMID 31217091

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort X | Cohort Y | Cohort A | Cohort B | Cohort C | Cohort D
Started | 10 | 17 | 0 | 0 | 0 | 0
Completed | 10 | 17 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Number of participants analyzed for Cohorts A-D is zero because no subjects were enrolled in Cohorts A-D because study was suspended due to lack of funding.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort X | Cohort Y | Cohort A | Cohort B | Cohort C | Cohort D | Total
Number analyzed (Participants) | 10 | 17 | 0 | 0 | 0 | 0 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 11 | 0 | 0 | 0 | 0 | 15
  >=65 years | 6 | 6 | 0 | 0 | 0 | 0 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 0 | 0 | 0 | 0 | 13
  Male | 5 | 9 | 0 | 0 | 0 | 0 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 10 | 16 | 0 | 0 | 0 | 0 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 5 | 0 | 0 | 0 | 0 | 6
  White | 9 | 12 | 0 | 0 | 0 | 0 | 21
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Primary Endpoint: Area Under the Curve (AUC), Sensitivity, and Specificity of VCI When Compared Against Standard of Care Imaging.
Description: The primary endpoint for both Phase 1 and Phase 2 of the study is to measure the AUC, Sensitivity, and Specificity of Velocity Curvature Index (VCI) when compared against standard of care CTA imaging for large vessel occlusion assessment. Initial assessment of outcome will be done after 18 months of study start and complete assessment will be done at the end of study's Phase 2.
Time Frame: 1 day
Population: It was pre-specified in "Outcome Measure Description" to report primary endpoint data for Phases 1 and 2 only, which includes subject Cohorts A-D. Phases 1 and 2 were never started due to lack of funding and no data was collected for subjects in Cohorts A-D that would allow data analysis regarding primary and secondary outcome measures.
Arm/Group | Cohort X | Cohort Y | Cohort A | Cohort B | Cohort C | Cohort D
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 day
Description: Device and procedure related adverse events collected only
Arm/Group | Cohort X | Cohort Y | Cohort A | Cohort B | Cohort C | Cohort D
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/17 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/17 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/10 | 0/17 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT05547412/Prot_SAP_000.pdf